CLINICAL TRIAL: NCT02305862
Title: An Open-label, Single-centre Randomized Study Evaluating the Effect of Treatment With Rosuvastatin 5/20mg on Atherosclerotic Disease as Measured by High-Resolution Contrast Enhanced Magnetic Resonance Imaging in Patients With Coronary Artery Disease and Hyperlipideimia
Brief Title: A High-Resolution Magnetic Resonance Imaging Study to Evaluate the Effect of Rosuvastatin on Carotid Atherosclerotic Plaques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Buxing Chen, Director of department of cardiology, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMARIROCAP
Record Dates: First submitted 2014-11-26; First posted 2014-12-03 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Arteriosclerosis; Diabetes Mellitus; Lipid Disorder
Keywords: Coronary Arteriosclerosis; Carotid Atherosclerotic Plaque; Rosuvastatin
MeSH Terms: conditions — Arteriosclerosis; Diabetes Mellitus; Lipid Metabolism Disorders; Coronary Artery Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low dose group (5mg) (Experimental): low dose Rosuvastatin
  Interventions: Drug: Rosuvastatin 5mg
- high dose group (20mg) (Experimental): high dose Rosuvastatin
  Interventions: Drug: Rosuvastatin 20mg

INTERVENTIONS:
Drug: Rosuvastatin 5mg — drug intervention
  Arms: low dose group (5mg)
Drug: Rosuvastatin 20mg — drug intervention
  Arms: high dose group (20mg)

SUMMARY:
The aim of this study is to assess whether high intensive statin therapy could regress carotid atherosclerotic plaques as determined by High-Resolution Contrast Enhanced Magnetic Resonance imaging (CE-MRI).

Enrolled patients have a baseline CE-MRI examination for screening carotid atherosclerotic plaques and are randomized to either low dose of Rosuvastatin (5mg) group or high dose of Rosuvastatin (20mg) group. After 26 weeks, all patients received CE-MRI examination again and each pair of baseline and follow-up CE-MRI assessments was analyzed in a blinded fashion. Moreover, lipid level and major adverse cardiovascular events are also evaluated during follow-up.

ELIGIBILITY:
Inclusion Criteria:

-Patients with coronary artery disease or carotid atherosclerotic plaque or hyperlipideimia or old myocardial infarction

Exclusion Criteria:

* Planning coronary stenting
* Heart failure
* Uncontrolled hypertension（≥200/110mmHg)
* Uncontrolled diabetes mellitus (HbA1C≥9.5%)
* Hepatic insufficiency
* Renal dysfunction
* Cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether 26 weeks of treatment with 5/20mg rosuvastatin results in regression of carotid atherosclerotic plaques as measured by CE-MRI | 26 weeks

SECONDARY OUTCOMES:
major adverse cardiovascular events | 26 weeks
To evaluate the change in lipid and lipoprotein levels as assessed by percentage change from baseline. | 26 weeks
To evaluate the change from baseline in liver function (AST/ALT) at 26 weeks | 26 weeks
To evaluate the change from baseline in renal function (serum creatine) at 26 weeks | 26 weeks
To evaluate the change from baseline in creatine kinase at 26 weeks | 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China